CLINICAL TRIAL: NCT04770675
Title: A Prospective, Multicenter, Post Market Study to Collect Data for Software Recognizing the Anatomical Structures as Well as Abnormalities in the Lung During a Bronchoscopy.
Brief Title: Post Market Study to Collect Data for Software Recognizing the Anatomical Structures During Bronchoscopy.
Status: Completed | Type: Observational
Sponsor: Qmed Consulting A/S (Industry)
Collaborators: Ambu A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: CIS-20
Record Dates: First submitted 2021-02-12; First posted 2021-02-25 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Tumor; Hemoptysis; Pulmonary Disease
Keywords: bronchoscope
MeSH Terms: conditions — Neoplasms; Hemoptysis; Lung Diseases | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment group: Any subject who is scheduled to undergo bronchoscopy as per routine clinical practice
  Interventions: Diagnostic Test: Bronchoscopy

INTERVENTIONS:
Diagnostic Test: Bronchoscopy — All subjects who are scheduled for a bronchoscopy may be eligible.

SUMMARY:
The primary aim is to develop a software algorithm that has the capacity to detect the normal 18 anatomical structures of the lung by using the position of the scope during the bronchoscopy procedure and using existing bronchoscopy technology.

DETAILED DESCRIPTION:
2.000 subjects, preferable 150-200 number of patients per site. The 2.000 videos will be divided into an 80%/20% split (training and testing). It is a wish to obtain a spread of videos coming from across Europe, preferable from Germany, France and Denmark, with up to 800 videos coming from Denmark

The patient population indicated are patients indicated for full airway bronchoscopy. Of this group it is the aim to enrol the following:

1. Patients with obstructing tumors (when tumor blocks the view of the camera) - no more than 5% (120 patients) of studies
2. Bronchoscopies on indication of haemoptysis (active bleeding) - no more than 5% (120 patients) of studies
3. Patients with stents or valves - no more than 5% (120 patients) of studies bronchoscopies.
4. Patients with former lung operations, partial or full resections - no more than 2% (48 patients).

ELIGIBILITY:
Inclusion Criteria:

1. Oral and written participant information has been given (NA for Denmark)
2. The subject has signed informed consent (NA for Denmark)
3. Patients indicated for full airway bronchoscopy (identifying all 18 anatomical segments)
4. Patients older than 18

Exclusion Criteria:

1. Subject with serious lung disease which investigator considers not appropriate for this examination.
2. Lack of patient cooperation for bronchoscopy (patient with mental disorders, dysgnosia, psychological disorder…)
3. Subjects unable to give consent (NA for Denmark)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The bronchoscope is used to confirm or exclude a diagnosis in adult patients with airway complaints to identify a potential disease.
Sampling Method: Probability Sample
Enrollment: 833 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of anatomical segments accessed during bronchoscopy | 1 day
  accurate photo documentation of all 18 anatomical segments +/- abnormalities

SECONDARY OUTCOMES:
Number of anatomical segments identified | 1 day
  Identified anatomical segments by the core lab/ Identified anatomical segments by the Machine Learning (after training, using the test videos).
Rate of total number of lesions detected | 1 day
  total lesions detected by the core lab/ total lesions detected by Machine Learning (after training, using the test videos).
Number of sections and lesions detected by core lab and machine learning | 1 day
  Anatomical sections + lesions detected by core lab versus anatomical sections + lesions detected by machine learning

CONTACTS AND LOCATIONS:
Overall Officials: Michael Perch, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Provide data to Ambu A/S that can not be identified without the identification log.
Supporting Information: Study Protocol, CSR
Time Frame: 2 years after study end
Access Criteria: restricted access with user accounts to electronic data capture system